CLINICAL TRIAL: NCT05744791
Title: The Influence of a Planned Movement and Physical Activity Program on the Physiological and Psychology Parameters in a Pediatric Population
Brief Title: Active Play Intervention for Preschoolers
Acronym: Active Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Danielle D Wadsworth, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-217 MR 1009
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Exercise
Keywords: Preschoolers; Active Play; Teacher guided interventions
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Two preschools. One will be randomized to the intervention and one to the control group.
Who Masked: Participant
Masking Description: Preschool children will not be aware of which intervention they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Play Intervention (Experimental): Preschool teachers will be asked to implement two active play activities each preschool day, one indoors and one outdoors. This is in addition to the current outdoor free play of 30 minutes each day. Each activity is 10-15 minutes for a total of 20-30 minutes per day.
  Interventions: Behavioral: Active Play planned movement program
- Control (No Intervention): Preschool teachers will continue to implement their regular curriculum. This consists of one outdoor play opportunity for 30 minutes each day.

INTERVENTIONS:
Behavioral: Active Play planned movement program — Teachers will implement an addition two physical activity opportunities that incorporate active play each day for a potential dose of 20-30 minutes per day and 100-150 minutes per week.
  Arms: Active Play Intervention

SUMMARY:
The goal of this randomized clinical trial is to examine the effects of a planned movement in preschool-aged children. The main question is to determine

* What are the effects of a planned movement program on physical activity, body composition, fundamental motor skills, and time on task in preschool children aged 3-5 years?

Researchers will compare a planned movement program to a control group, where current instruction is implemented.

DETAILED DESCRIPTION:
A majority of preschool children do not participate in the recommended levels of physical activity and are deficient in fundamental motor skills. These deficits may also impact body composition. Preschool teachers serve as the gateway to providing physical activity opportunities at preschool but many fail to do so. As play is developmentally appropriate for preschools and part of many curriculums adding active elements to play may be a feasible solution for teachers to implement physical activity opportunities. This project will evaluate the effect of a planned movement program that incorporates elements of active play on preschoolers' body composition, physical activity, time on task, and fundamental motor skills at week 0, week 12, and week 24. Physical Activity will be assessed throughout the school year with a wrist-worn wearable accelerometer. Body composition will be assessed with a foot-to-foot bioelectrical impedance scale. Fundamental motor skills will be assessed by the Peabody Developmental Motor Scales 2nd Edition and Time on-task will be measured by observing children in their classroom. The outcomes of this study will be used to implement sustainable physical activity programming for preschoolers.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 5 years of age
* attending one of the preschools 5 days a week.

Exclusion Criteria:

* less than 3 years of age
* greater than 5 years of age at the beginning of the study
* attends the preschool 2 days or 3 days a week

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 12 weeks
  An accelerometer attached at the wrist will measure physical activity over 24 hours for 5 days at baseline and 12 weeks
Body composition | 12 weeks
  Percent body fat, ratio of fat mass to lean mass, will be assessed with electrical impedance.
Fundamental motor skills | 12 weeks
  The fundamental motor skill gross quotient will be measured with the Peabody Developmental Motor Scales, Second Edition 2nd edition (PDMS-2). The sum of points comprises the raw scores for each subscale. Raw scores range for each subscale are 6-60 for Stationary Skills, 6-178 for Locomotion Skills, and 6-48 for Object Manipulation Skills. Using age-appropriate tables in the testing manual, we will convert the raw scores to standardized scores (0-20) and summed them to determine the gross motor quartile (GMQ), which has a range of 41 - 164. A higher score indicates a more favorable outcome.
Time on Task | 12 weeks
  The percentage of time spent on task will be observed and presented as a ratio of time on task to time spent off task.

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States